CLINICAL TRIAL: NCT03842163
Title: PREVALENCE AND CHARACTERISTICS OF TRANSTHYRETIN AMYLOIDOSIS IN PATIENTS WITH LEFT VENTRICULAR HYPERTROPHY OF UNKNOWN ETIOLOGY TTRACK
Brief Title: Prevalence and Characteristics of Transthyretin Amyloidosis in Patients With Left Ventricular Hypertrophy of Unknown Etiology
Acronym: TTRACK
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B3461058; TTRACK (Other: Alias Study Number)
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Results first posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2023-05

CONDITIONS: Transthyretin Amyloidosis Cardiomyopathy (ATTR-CM)
Keywords: Scintigraphy; Gammagraphy; TTR; ATTR; Hypertrophic cardiomyopathy (HCM); HCM
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with LVH of unknown etiology
  Interventions: Diagnostic Test: Diagnosis of TTR amyloidosis cardiomyopathy

INTERVENTIONS:
Diagnostic Test: Diagnosis of TTR amyloidosis cardiomyopathy — Diagnosis of TTR amyloidosis cardiomyopathy with scintigraphy

SUMMARY:
The main purpose of this study is to determine the prevalence of ATTR Cardiomyopathy among patients admitted due to Left Ventricular Hypertrophy (LVH) >15mm of unknown etiology by using a 99mTc-tracer scintigraphy based protocol

ELIGIBILITY:
Inclusion criteria:

* Patient signed inform consent.
* Males and Females.
* Age ≥50 years.
* Left ventricular hypertrophy (LVH) defined as end-diastolic LV maximum wall thickness (MWT) ≥15mm in Echocardiogram.
* Plan to undergo or recently underwent radionuclide bone scintigraphy and/or SPECT with any of the following radio labelled tracers: 99mTc-DPD or 99mTc-PYP or 99mTc-HMDP.

Exclusion criteria:

* Etiological diagnosis explaining the LVH (p.e. Sarcomeric HCM, Myeloma, Fabry disease, Sarcoidosis, Any type of amyloidosis (AA, AL, TTR)
* Severe aortic stenosis defined as aortic valve area (AVA) < 1.0 cm2

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HCM from undiagnosed etiology
Sampling Method: Non-Probability Sample
Enrollment: 812 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- Australia (2):
  - The Prince Charles Hospital, Chermside
  - The Alfred Department of Cardiology, Melbourne
- Medizinische Universität Innsbruck - Universitätsklinik für Innere Medizin III, Kardiologie, Innsbruck, Austria
- France (4):
  - Centre Hospitalier Universitaire de Caen, Caen, Cedex
  - Hopital Henri Mondor, Service de Pharmacologie Clinique, Créteil
  - CHU de Nantes, Nantes
  - CHU de Toulouse, Toulouse
- Italy (2):
  - Divisione di Cardiologia, Bologna
  - Careggi Hospital, Florence
- Portugal (2):
  - Centro Hospitalar e Universitario de Coimbra, Coimbra
  - Centro Hospitalar de Lisboa Central, E.P.E., Lisbon
- Romania (2):
  - Fundeni Clinical Institute, Bucharest
  - Inherited Cardiovascular Diseases - Cardiology Institute, Bucharest
- East Slovak Institute of Cardiovascular Diseases, Košice, Slovakia
- University Medical Centre Ljubljana - Department of Cardiology, Ljubljana, Slovenia
- Spain (2):
  - Cardiomyopathy Unit, Department of Cardiology, Majadahonda, Madrid
  - Hospital Universitario A Coruna, A Coruña
- The Heart Hospital - University College London Hospitals Nhs Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Garcia-Pavia P, Del Moral FJH, Cappelli F, Piriou N, Barriales-Villa R, Munteanu C, Bahus C, Keohane D, Mallaina P, Itti E, Damy T, Elliott P. Nuclear imaging and echocardiographic findings in hypertrophic cardiomyopathy with and without ATTR-CM. ESC Heart Fail. 2025 Dec;12(6):4349-4358. doi: 10.1002/ehf2.15440. Epub 2025 Oct 13. PMID 41081448
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3461058

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants diagnosed with left ventricular hypertrophy (LVH) confirmed by bone scintigraphy and/or single photon emission computed tomography (SPECT) and greater than or equal to (>=) 50 years of age were observed in this study.
Pre-assignment Details: Data from eligible participants were retrieved and observed from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years).
Groups:
- All Participants: Participants diagnosed with LVH of unknown etiology confirmed by bone scintigraphy and/or SPECT were included.
Period: Overall Study
Arm/Group | All Participants
Started | 812
Full Analysis Set 1 | 766
Full Analysis Set 2 (Subset of FAS 1) | 245
Full Analysis Set 3 (Subset of FAS 2) | 208
Full Analysis Set 3.1 | 137
Full Analysis Set 3.2 | 56
Completed | 766
Not Completed | 46
Not completed — Did not meet inclusion criteria (age less than 50 years) | 2
Not completed — Scintigraphy was not performed | 44

BASELINE CHARACTERISTICS:
Population: Full Analysis Set 1 (FAS1) included all participants who met eligibility criteria and with a radionuclide bone scintigraphy and/or SPECT performed with 99mTechnetium-3,3-diphosphono-1,2-propanodi-carboxylic acid (99mTc-DPD) or 99mTechnetium-pyrophosphate (99mTc-PYP) or 99mTechnetium-hydroxymethylene diphosphonate (99mTc-HMDP).
Arm/Group | All Participants
Number analyzed (Participants) | 766
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233
  Male | 533
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 665
  Caucasian & Portuguese (or Portuguese parents) | 47
  African | 21
  Asian | 27
  Other | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Cardiac Fixation at the Radionuclide Bone Scintigraphy and/or Single Photon Emission Computed Tomography (SPECT): FAS1
Description: Percentage of participants with cardiac fixation on a radionuclide bone scintigraphy and/or SPECT performed with 99mTc-DPD or 99mTc-PYP or 999mTc-HMDP among participants with LVH from an undiagnosed etiology were reported in this outcome measure. Scintigraphy was defined at each bone site according to the standard grading: Grade 0 = absent cardiac uptake, Grade 1=mild uptake less than bone, Grade 2=moderate uptake equal to bone and Grade 3=high uptake greater than bone.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS1 included all participants who met eligibility criteria and with a radionuclide bone scintigraphy and/or SPECT performed with 99mTc-DPD/99mTc-PYP/99mTc-HMDP.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 766
Percentage of participants | 32.0 [28.8 to 35.4]

2. Secondary Outcome: Percentage of Participants With Transthyretin Amyloid (ATTR): FAS 1
Description: Transthyretin amyloidosis is a slowly progressive condition characterized by the buildup of abnormal deposits of a protein called amyloid (amyloidosis) in the body's organs and tissues.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS 1 included all participants who met eligibility criteria and with a radionuclide bone scintigraphy and/or SPECT performed with 99mTc-DPD/99mTc-PYP/99mTc-HMDP.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 766
Percentage of participants | 17.9 [15.3 to 20.8]

3. Secondary Outcome: Percentage of Participants With ATTR or With Suspicion of Monoclonal Gammopathy of Undetermined Significance (MGUS) / Light Chain Amyloidosis (AL): FAS 1
Description: as for outcome 2
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 766
Percentage of participants | 25.2 [22.3 to 28.4]

4. Secondary Outcome: Percentage of Participants With Hereditary Transthyretin Amyloid (ATTRv): Full Analysis Set 2 (FAS 2)
Description: Percentage of participants with hereditary ATTRv were reported in this outcome measure. ATTR participants with a ATTR gene sequencing with variant transthyretin was considered as ATTRv.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS 2 included all eligible participants with a radionuclide bone scintigraphy and/or SPECT performed with 99mTc-DPD/99mTc-PYP/99mTc-HMDP and with grading of cardiac retention equal to grade 1, grade 2 or grade 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 245
Percentage of participants | 6.5 [3.8 to 10.8]

5. Secondary Outcome: Percentage of Participants With Hereditary Transthyretin Amyloid (ATTRv): Full Analysis Set 3 (FAS 3)
Description: as for outcome 4
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS 3 included all eligible participants with radionuclide bone scintigraphy and/or SPECT performed with 99mTc-DPD/99mTc-PYP/99mTc-HMDP and with grading of cardiac retention equal to grade 2 or grade 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 208
Percentage of participants | 6.9 [4.1 to 11.5]

6. Secondary Outcome: Percentage of Participants With Hereditary Transthyretin Amyloid (ATTRv): FAS 3.1
Description: as for outcome 4
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS 3.1 included all eligible participants with grade 2-3 without monoclonal protein abnormalities (ATTR amyloidosis).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 137
Percentage of participants | 8.7 [4.9 to 14.8]

7. Secondary Outcome: Percentage of Participants With Hereditary Transthyretin Amyloid (ATTRv): FAS 3.2
Description: as for outcome 4
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS 3.2 included all eligible participants with grade 2-3 with monoclonal protein abnormalities (undefined etiology, cardiac ATTR amyloidosis, or MGUS or AL amyloidosis).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 56
Percentage of participants | 3.7 [1.0 to 12.5]

8. Secondary Outcome: Percentage of Participants With Wild Type Transthyretin Amyloid (ATTRwt): FAS 2
Description: Percentage of participants with ATTRwt were reported in this outcome measure. ATTR participants with a ATTR gene sequencing with a result of 'no mutation' was considered as ATTRwt.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 245
Percentage of participants | 93.5 [89.2 to 96.2]

9. Secondary Outcome: Percentage of Participants With Wild Type Transthyretin Amyloid (ATTRwt): FAS 3
Description: as for outcome 8
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 208
Percentage of participants | 93.1 [88.5 to 95.9]

10. Secondary Outcome: Percentage of Participants With Wild Type Transthyretin Amyloid (ATTRwt): FAS 3.1
Description: as for outcome 8
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS 3.1 included all eligible participants with grade 2-3 without monoclonal protein abnormalities (ATTR amyloidosis).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 137
Percentage of participants | 91.3 [85.2 to 95.1]

11. Secondary Outcome: Percentage of Participants With Wild Type Transthyretin Amyloid (ATTRwt): FAS 3.2
Description: as for outcome 8
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 56
Percentage of participants | 96.3 [87.5 to 99.0]

12. Secondary Outcome: Number of Participants With Transthyretin (TTR) Genetic Mutations Among Those Who Had Positive Scintigraphy: FAS 2
Description: Scintigraphy is the procedure used to diagnose, stage, and monitor disease. A small amount of a radioactive chemical (radionuclide) was injected into a vein or swallowed. Number of participants with TTR genetic mutations among those who had positive scintigraphy were reported in this outcome measure.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS 2 included all eligible participants with a radionuclide bone scintigraphy and/or SPECT performed with 99mTc-DPD/99mTc-PYP/99mTc-HMDP and with grading of cardiac retention equal to grade 1, grade 2 or grade 3. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 200
Participants | 13

13. Secondary Outcome: Number of Participants With Transthyretin (TTR) Genetic Mutations Among Those Who Had Positive Scintigraphy: FAS 3
Description: as for outcome 12
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 208
Participants | 13

14. Secondary Outcome: Number of Participants With Transthyretin (TTR) Genetic Mutations Among Those Who Had Positive Scintigraphy: FAS 3.1
Description: as for outcome 12
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS 3.1 included all eligible participants with grade 2-3 without monoclonal protein abnormalities (ATTR amyloidosis). Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 127
Participants | 11

15. Secondary Outcome: Number of Participants With Transthyretin (TTR) Genetic Mutations Among Those Who Had Positive Scintigraphy: FAS 3.2
Description: as for outcome 12
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS 3.2 included all eligible participants with grade 2-3 with monoclonal protein abnormalities (undefined etiology, cardiac ATTR amyloidosis, or MGUS or AL amyloidosis). Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 54
Participants | 2

16. Secondary Outcome: Percentage of Participants With Any Familial History of Known Cardiomyopathy (CM), Polyneuropathy (PN) or Sudden Cardiac Death (SCD) Among Their Relatives (Parents, Siblings and 2nd /3rd Grade Family): FAS 1
Description: Percentage of participants with any of the familial history of known CM, PN or SCD among their relatives were reported in this outcome measure. Family history for each disease was considered for 1st degree parent, siblings, and 2nd/3rd grade family. CM was defined by the presence of a left ventricular (LV) wall thickness greater than or equal to (>=) 15 mm in one or more LV myocardial segments that is not explained solely by abnormal loading conditions. Polyneuropathy was defined as the simultaneous malfunction of many peripheral nerves throughout the body. SCD was defined as death due to a cardiovascular cause that occurs within one hour of the onset of symptoms. A sudden cardiac arrest occurs when the heart stops beating or is not beating sufficiently to maintain perfusion and life.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 766
Percentage of participants | 17.1 [14.6 to 19.9]

17. Secondary Outcome: Percentage of Participants With Any Familial History of Known Cardiomyopathy (CM), Polyneuropathy (PN) or Sudden Cardiac Death (SCD) Among Their Relatives (Parents, Siblings and 2nd /3rd Grade Family): FAS 2
Description: Percentage of participants with any of the familial history of known CM, PN or SCD among their relatives were reported in this outcome measure. Family history for each disease was considered for 1st degree parent, siblings, and 2nd/3rd grade family. CM was defined by the presence of a LV wall thickness >= 15 mm in one or more LV myocardial segments that is not explained solely by abnormal loading conditions. Polyneuropathy was defined as the simultaneous malfunction of many peripheral nerves throughout the body. SCD was defined as death due to a cardiovascular cause that occurs within one hour of the onset of symptoms. A sudden cardiac arrest occurs when the heart stops beating or is not beating sufficiently to maintain perfusion and life.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 245
Percentage of participants | 11.8 [8.4 to 16.5]

18. Secondary Outcome: Percentage of Participants With Any Familial History of Known Cardiomyopathy (CM), Polyneuropathy (PN) or Sudden Cardiac Death (SCD) Among Their Relatives (Parents, Siblings and 2nd /3rd Grade Family): FAS 3
Description: as for outcome 17
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 208
Percentage of participants | 9.6 [6.3 to 14.4]

19. Secondary Outcome: Percentage of Participants With Any Familial History of Known Cardiomyopathy (CM), Polyneuropathy (PN) or Sudden Cardiac Death (SCD) Among Their Relatives (Parents, Siblings and 2nd /3rd Grade Family): FAS 3.1
Description: as for outcome 17
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS 3.1 included all eligible participants with grade 2-3 without monoclonal protein abnormalities (ATTR amyloidosis).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 137
Percentage of participants | 10.9 [6.7 to 17.3]

20. Secondary Outcome: Percentage of Participants With Any Familial History of Known Cardiomyopathy (CM), Polyneuropathy (PN) or Sudden Cardiac Death (SCD) Among Their Relatives (Parents, Siblings and 2nd /3rd Grade Family): FAS 3.2
Description: as for outcome 17
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 56
Percentage of participants | 7.1 [2.8 to 17.0]

21. Secondary Outcome: Percentage of Participants With Senso-Motor Polyneuropathy: FAS 2
Description: Participants with at least one red flag in the neurological part of the ATTR-Amyloidosis red flags Electronic Case Report Form (e-CRF) part was considered as participants with a senso-motor polyneuropathy.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 245
Percentage of participants | 80.0 [74.5 to 84.5]

22. Secondary Outcome: Percentage of Participants With Senso-Motor Polyneuropathy: FAS 3
Description: Participants with at least one red flag in the neurological part of the ATTR-Amyloidosis red flags e-CRF part was considered as participants with a senso-motor polyneuropathy.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 208
Percentage of participants | 86.1 [80.7 to 90.1]

23. Secondary Outcome: Percentage of Participants With Senso-Motor Polyneuropathy: FAS 3.1
Description: as for outcome 22
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS 3.1 included all eligible participants with grade 2-3 without monoclonal protein abnormalities (ATTR amyloidosis).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 137
Percentage of participants | 89.8 [83.6 to 93.8]

24. Secondary Outcome: Percentage of Participants With Senso-Motor Polyneuropathy: FAS 3.2
Description: as for outcome 22
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 56
Percentage of participants | 85.7 [74.3 to 92.6]

25. Secondary Outcome: Percentage of Participants With Carpal Tunnel Syndrome (CTS): FAS 2
Description: CTS was defined as a common neurological disorder that occurs when the median nerve, which runs from your forearm into the palm of the hand, becomes pressed or squeezed at the wrist. Participants with a CTS were participants with a bilateral or unilateral CTS.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 245
Percentage of participants | 48.6 [42.4 to 54.8]

26. Secondary Outcome: Percentage of Participants With Carpal Tunnel Syndrome (CTS): FAS 3
Description: as for outcome 25
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 208
Percentage of participants | 54.8 [48.0 to 61.4]

27. Secondary Outcome: Percentage of Participants With Carpal Tunnel Syndrome (CTS): FAS 3.1
Description: as for outcome 25
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS 3.1 included all eligible participants with grade 2-3 without monoclonal protein abnormalities (ATTR amyloidosis).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 137
Percentage of participants | 60.6 [52.2 to 68.4]

28. Secondary Outcome: Percentage of Participants With Carpal Tunnel Syndrome (CTS): FAS 3.2
Description: as for outcome 25
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 56
Percentage of participants | 48.2 [35.7 to 61.0]

29. Secondary Outcome: Percentage of Participants With Autonomic Dysfunction: FAS 2
Description: Participants with autonomic dysfunction were participants with at least one autonomic sign or autonomic symptom = "Yes".
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 245
Percentage of participants | 55.9 [49.7 to 62.0]

30. Secondary Outcome: Percentage of Participants With Autonomic Dysfunction: FAS 3
Description: Participants with autonomic dysfunction were participants with at least one autonomic sign or autonomic symptom = "Yes".
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 208
Percentage of participants | 58.7 [51.9 to 65.1]

31. Secondary Outcome: Percentage of Participants With Autonomic Dysfunction: FAS 3.1
Description: Participants with autonomic dysfunction were participants with at least one autonomic sign or autonomic symptom = "Yes".
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS 3.1 included all eligible participants with grade 2-3 without monoclonal protein abnormalities (ATTR amyloidosis).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 137
Percentage of participants | 61.3 [53.0 to 69.1]

32. Secondary Outcome: Percentage of Participants With Autonomic Dysfunction: FAS 3.2
Description: Participants with autonomic dysfunction were participants with at least one autonomic sign or autonomic symptom = "Yes".
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 56
Percentage of participants | 57.1 [44.1 to 69.2]

33. Secondary Outcome: Percentage of Participants With Cardiological Manifestations: FAS 2
Description: Participants with cardiological manifestations was defined as participants with at least one of the following criteria fulfilled from data collected from e-CRF: cardiological assessments: atrial fibrillation (yes permanent), pacemaker (yes), AICD (yes); in magnetic resonance imaging (MRI) part: LGE (positive); electrocardiogram (ECG) part: PR interval less than (<) 80 milliseconds (ms) or greater than (>) 350 ms QRS interval < 60 ms or > 250 ms, Sokolow index < 1 mm or > 70 mm, pseudo MI pattern (yes), PPOr precordial R wave progression(yes), LBBB, RBBB, paced and intraventricular conduct delay (ticked), LVOT (yes), if longitudinal strain is done, strain apical preserved (yes), LV end-diastolic diameter <20 mm or >80 mm, MWT <15 mm or >100 mm, MWT at septum <3 mm or >50 mm, MWT posterior wall <3 mm or >50 mm, LV mass index <40 g/m^2 or >160 g/m^2, Maximal aortic velocity >5 m/s, Mean gradient of Aortic valvular stenosis >70 mmHg, Area of Aortic valvular stenosis <0.2 cm^2 or >3 cm^2.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 245
Percentage of participants | 98.0 [95.3 to 99.1]

34. Secondary Outcome: Percentage of Participants With Cardiological Manifestations: FAS 3
Description: Participants with cardiological manifestations was defined as participants with at least one of the following criteria fulfilled from data collected from e-CRF: cardiological assessments: atrial fibrillation (yes permanent), pacemaker (yes), AICD (yes); in magnetic resonance imaging (MRI) part: LGE (positive); electrocardiogram (ECG) part: PR interval < 80 ms or > 350 ms QRS interval < 60 ms or > 250 ms, Sokolow index < 1 mm or > 70 mm, pseudo MI pattern (yes), PPOr precordial R wave progression(yes), LBBB, RBBB, paced and intraventricular conduct delay (ticked), LVOT (yes), if longitudinal strain is done, strain apical preserved (yes), LV end-diastolic diameter <20 mm or >80 mm, MWT <15 mm or >100 mm, MWT at septum <3 mm or >50 mm, MWT posterior wall <3 mm or >50 mm, LV mass index <40 g/m^2 or >160 g/m^2, Maximal aortic velocity >5 m/s, Mean gradient of Aortic valvular stenosis >70 mmHg, Area of Aortic valvular stenosis <0.2 cm^2 or >3 cm^2.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 208
Percentage of participants | 98.1 [95.2 to 99.2]

35. Secondary Outcome: Percentage of Participants With Cardiological Manifestations: FAS 3.1
Description: as for outcome 34
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS 3.1 included all eligible participants with grade 2-3 without monoclonal protein abnormalities (ATTR amyloidosis).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 137
Percentage of participants | 97.8 [93.8 to 99.3]

36. Secondary Outcome: Percentage of Participants With Cardiological Manifestations: FAS 3.2
Description: as for outcome 34
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 56
Percentage of participants | 98.2 [90.6 to 99.7]

37. Secondary Outcome: Percentage of Participants With Laboratory Abnormalities: FAS 2
Description: Laboratory parameters that were considered as out of range included creatinine <45 micromole per liter (μmol/L) or greater than 104 μmol/L w; haemoglobin, participants with a value lower than 11.5 grams per deciliter (g/dL) or higher than 16 g/dL was considered as out of range; Brain natriuretic peptide (BNP) value higher than 100 picograms per milliliter (pg/mL); N-terminal pro-brain natriuretic peptide (NTproBNP), value higher than 125 pg/mL; Troponin I value higher than 26 pg/mL.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 245
Percentage of participants
  Creatinine out of range | 37.6 [31.7 to 43.8]
  Haemoglobin out of range | 30.2 [24.8 to 36.2]
  BNP out of range | 62.9 [56.7 to 68.7]
  NTproBNP out of range | 81.2 [75.9 to 85.6]
  Troponin I out of range | 3.7 [1.9 to 6.8]

38. Secondary Outcome: Percentage of Participants With Laboratory Abnormalities: FAS 3
Description: Laboratory parameters that were considered as out of range included creatinine <45 μmol/L or greater than 104 μmol/L w; haemoglobin value lower than 11.5 g/dL or higher than 16 g/dL was considered as out of range; Brain natriuretic peptide (BNP) value higher than 100 pg/mL; N-terminal pro-brain natriuretic peptide (NTproBNP), value higher than 125 pg/mL; Troponin I value higher than 26 pg/mL.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 208
Percentage of participants
  Creatinine out of range | 42.3 [35.8 to 49.1]
  Haemoglobin out of range | 33.2 [27.1 to 39.8]
  BNP out of range | 69.7 [63.2 to 75.6]
  NTproBNP out of range | 88.9 [84.0 to 92.5]
  Troponin I out of range | 3.8 [2.0 to 7.4]

39. Secondary Outcome: Percentage of Participants With Laboratory Abnormalities: FAS 3.1
Description: as for outcome 38
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS 3.1 included all eligible participants with grade 2-3 without monoclonal protein abnormalities (ATTR amyloidosis).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 137
Percentage of participants
  Creatinine out of range | 34.3 [26.9 to 42.6]
  Haemoglobin out of range | 34.3 [26.9 to 42.6]
  BNP out of range | 68.6 [60.4 to 75.8]
  NTproBNP out of range | 90.5 [84.4 to 94.4]
  Troponin I out of range | 4.4 [2.0 to 9.2]

40. Secondary Outcome: Percentage of Participants With Laboratory Abnormalities: FAS 3.2
Description: as for outcome 38
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 56
Percentage of participants
  Creatinine out of range | 58.9 [45.9 to 70.8]
  Haemoglobin out of range | 35.7 [24.5 to 48.8]
  BNP out of range | 89.3 [78.5 to 95.0]
  NTproBNP out of range | 98.2 [90.6 to 99.7]
  Troponin I out of range | 1.8 [0.3 to 9.4]

41. Secondary Outcome: Number of Participants According to Presence of Neurological Red Flag: FAS1
Description: Participants were classified according to presence of neurological red flag as 'Yes' or 'No'.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 766
Participants
  Yes | 143
  No | 623

42. Secondary Outcome: Number of Participants According to Presence of Neurological Red Flag: FAS 2
Description: Participants were classified according to presence of neurological red flag as 'Yes' or 'No'.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 245
Participants
  Yes | 142
  No | 103

43. Secondary Outcome: Number of Participants According to Discrepancies Between Scintigraphy Result and Single Photon Emission Computed Tomography (SPECT) Result: FAS1
Description: Grade of scintigraphy evaluated by the investigator and Grade of SPECT: Grade 0 = absent cardiac uptake, Grade 1=mild uptake less than bone, Grade 2=moderate uptake equal to bone and Grade 3=high uptake greater than bone. Only categories with non-zero values were reported.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS1 included all participants who met eligibility criteria and with a radionuclide bone scintigraphy and/or SPECT performed with 99mTc-DPD/99mTc-PYP/99mTc-HMDP. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 75
Participants
  Investigator: Grade 0; SPECT: Grade 0 | 43
  Investigator: Grade 0; SPECT: Grade 1 | 3
  Investigator: Grade 1; SPECT: Grade 1 | 5
  Investigator: Grade 2; SPECT: Grade 2 | 16
  Investigator: Grade 3; SPECT: Grade 3 | 8

44. Secondary Outcome: Cardiological Assessments - Blood Pressure: FAS 2
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were evaluated.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Participants
Number analyzed (Participants) | 238
mmHg
  DBP | 75.6 (12.4)
  SBP | 132.5 (20.0)

45. Secondary Outcome: Cardiological Assessments - Blood Pressure: FAS 3
Description: SBP and DBP were evaluated.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS 3 included all eligible participants with radionuclide bone scintigraphy and/or SPECT performed with 99mTc-DPD/99mTc-PYP/99mTc-HMDP and with grading of cardiac retention equal to grade 2 or grade 3. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Participants
Number analyzed (Participants) | 203
mmHg
  DBP | 74.6 (12.0)
  SBP | 131.0 (19.0)

46. Secondary Outcome: Cardiological Assessments - Blood Pressure: FAS 3.1
Description: SBP and DBP were evaluated.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Participants
Number analyzed (Participants) | 133
mmHg
  DBP | 75.6 (11.8)
  SBP | 130.9 (18.1)

47. Secondary Outcome: Cardiological Assessments - Blood Pressure: FAS 3.2
Description: SBP and DBP were evaluated.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Participants
Number analyzed (Participants) | 55
mmHg
  DBP | 74.2 (11.9)
  SBP | 131.9 (20.5)

48. Secondary Outcome: Number of Participants According to History of Clinical Parameters at Baseline: FAS 2
Description: Clinical parameters' assessment for hypertension, antihypertensive medication, coronary artery disease, renal insufficiency, diabetes mellitus, lumbar spinal stenosis, carpal tunnel syndrome was categorized as 'Yes' and 'No', where Yes indicated presence and No indicated absence.
Time Frame: Baseline
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 245
Participants
  Diagnosed hypertension: No | 78
  Diagnosed hypertension: Yes | 167
  Antihypertensive medication: No | 89
  Antihypertensive medication: Yes | 156
  Coronary artery disease: No | 184
  Coronary artery disease: Yes | 61
  Renal insufficiency: No | 177
  Renal insufficiency: Yes | 68
  Diabetes Mellitus: No | 193
  Diabetes Mellitus: Yes | 52
  Lumbar spinal stenosis: No | 221
  Lumbar spinal stenosis: Yes | 24
  Carpal tunnel syndrome: No | 164
  Carpal tunnel syndrome: Yes | 81

49. Secondary Outcome: Number of Participants According to History of Clinical Parameters at Baseline: FAS 3
Description: as for outcome 48
Time Frame: Baseline
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 208
Participants
  Diagnosed hypertension: No | 77
  Diagnosed hypertension: Yes | 131
  Antihypertensive medication: No | 88
  Antihypertensive medication: Yes | 120
  Coronary artery disease: No | 162
  Coronary artery disease: Yes | 46
  Renal insufficiency: No | 147
  Renal insufficiency: Yes | 61
  Diabetes Mellitus: No | 175
  Diabetes Mellitus: Yes | 33
  Lumbar spinal stenosis: No | 184
  Lumbar spinal stenosis: Yes | 24
  Carpal tunnel syndrome: No | 130
  Carpal tunnel syndrome: Yes | 78

50. Secondary Outcome: Number of Participants According to History of Clinical Parameters at Baseline: FAS 3.1
Description: as for outcome 48
Time Frame: Baseline
Population: FAS 3.1 included all eligible participants with grade 2-3 without monoclonal protein abnormalities (ATTR amyloidosis).
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 137
Participants
  Diagnosed hypertension: No | 49
  Diagnosed hypertension: Yes | 88
  Antihypertensive medication: No | 57
  Antihypertensive medication: Yes | 80
  Coronary artery disease: No | 112
  Coronary artery disease: Yes | 25
  Renal insufficiency: No | 102
  Renal insufficiency: Yes | 35
  Diabetes Mellitus: No | 118
  Diabetes Mellitus: Yes | 19
  Lumbar spinal stenosis: No | 121
  Lumbar spinal stenosis: Yes | 16
  Carpal tunnel syndrome: No | 80
  Carpal tunnel syndrome: Yes | 57

51. Secondary Outcome: Number of Participants According to History of Clinical Parameters at Baseline: FAS 3.2
Description: as for outcome 48
Time Frame: Baseline
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 56
Participants
  Diagnosed hypertension: No | 19
  Diagnosed hypertension: Yes | 37
  Antihypertensive medication: No | 22
  Antihypertensive medication: Yes | 34
  Coronary artery disease: No | 43
  Coronary artery disease: Yes | 13
  Renal insufficiency: No | 35
  Renal insufficiency: Yes | 21
  Diabetes Mellitus: No | 45
  Diabetes Mellitus: Yes | 11
  Lumbar spinal stenosis: No | 50
  Lumbar spinal stenosis: Yes | 6
  Carpal tunnel syndrome: No | 37
  Carpal tunnel syndrome: Yes | 19

52. Secondary Outcome: Number of Participants Classified According to New York Heart Association (NYHA) Class: FAS 2
Description: Participants classified according to NYHA class as Class I, Class II, Class III, Class IV were reported in this outcome measure. Class I: no symptoms and no limitation in ordinary physical activity, such as shortness of breath when walking, climbing stairs. Class II: mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity. Class III: marked limitation in activity due to symptoms, even during less-than-ordinary activity, such as walking short distances (20-100 meters), comfortable only at rest. Class IV: severe limitations and experienced symptoms even while at rest, mostly bedbound participants.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 245
Participants
  Class I | 50
  Class II | 130
  Class III | 57
  Class IV | 7
  Missing data | 1

53. Secondary Outcome: Number of Participants Classified According to New York Heart Association (NYHA) Class: FAS 3
Description: as for outcome 52
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 208
Participants
  Class I | 45
  Class II | 112
  Class III | 45
  Class IV | 5
  Missing data | 1

54. Secondary Outcome: Number of Participants Classified According to New York Heart Association (NYHA) Class: FAS 3.1
Description: as for outcome 52
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS 3.1 included all eligible participants with grade 2-3 without monoclonal protein abnormalities (ATTR amyloidosis).
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 137
Participants
  Class I | 34
  Class II | 69
  Class III | 30
  Class IV | 3
  Missing data | 1

55. Secondary Outcome: Number of Participants Classified According to New York Heart Association (NYHA) Class: FAS 3.2
Description: as for outcome 52
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 56
Participants
  Class I | 5
  Class II | 38
  Class III | 11
  Class IV | 2

56. Secondary Outcome: Number of Participants With Atrial Fibrillation Assessment: FAS 2
Description: Participants were classified according to presence of atrial fibrillation as 'No', 'Yes permanent', 'Yes in the past' and were reported in this outcome measure.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 245
Participants
  No | 120
  Yes permanent | 90
  Yes in the past | 35

57. Secondary Outcome: Number of Participants With Atrial Fibrillation Assessment: FAS 3
Description: as for outcome 56
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 208
Participants
  No | 105
  Yes permanent | 78
  Yes in the past | 25

58. Secondary Outcome: Number of Participants With Atrial Fibrillation Assessment: FAS 3.1
Description: as for outcome 56
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS 3.1 included all eligible participants with grade 2-3 without monoclonal protein abnormalities (ATTR amyloidosis).
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 137
Participants
  No | 65
  Yes permanent | 52
  Yes in the past | 20

59. Secondary Outcome: Number of Participants With Atrial Fibrillation Assessment: FAS 3.2
Description: as for outcome 56
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 56
Participants
  No | 28
  Yes permanent | 23
  Yes in the past | 5

60. Secondary Outcome: Number of Participants With Pacemaker and Implantable Cardiac Defibrillator (ICD): FAS 2
Description: Participants who used pacemaker and ICD were reported in this outcome measure.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 245
Participants
  Pacemaker: Yes | 30
  Pacemaker: No | 215
  ICD: Yes | 0
  ICD: No | 245

61. Secondary Outcome: Number of Participants With Pacemaker and Implantable Cardiac Defibrillator (ICD): FAS 3
Description: Participants who used pacemaker and ICD were reported in this outcome measure.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 208
Participants
  Pacemaker: Yes | 30
  Pacemaker: No | 178
  ICD: Yes | 0
  ICD: No | 208

62. Secondary Outcome: Number of Participants With Pacemaker and Implantable Cardiac Defibrillator (ICD): FAS 3.1
Description: Participants who used pacemaker and ICD were reported in this outcome measure.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: FAS 3.1 included all eligible participants with grade 2-3 without monoclonal protein abnormalities (ATTR amyloidosis).
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 137
Participants
  Pacemaker: Yes | 20
  Pacemaker: No | 117
  ICD: Yes | 0
  ICD: No | 137

63. Secondary Outcome: Number of Participants With Pacemaker and Implantable Cardiac Defibrillator (ICD): FAS 3.2
Description: Participants who used pacemaker and ICD were reported in this outcome measure.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 56
Participants
  Pacemaker: Yes | 7
  Pacemaker: No | 49
  ICD: Yes | 0
  ICD: No | 56

64. Secondary Outcome: Number of Participants With Magnetic Resonance Imaging (MRI) Scan Performed Using Late Gadolinium Enhancement (LGE): FAS 2
Description: Participants with MRI scan performed using LGE classified as 'negative' and 'positive' were reported in this outcome measure. LGE was defined as method where cardiovascular magnetic resonance (CMR) images were obtained after the administration of gadolinium contrast material that accumulated into a tissue with increased extra cellular space.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 66
Participants
  Negative | 11
  Positive | 55

65. Secondary Outcome: Number of Participants With Magnetic Resonance Imaging (MRI) Scan Performed Using Late Gadolinium Enhancement (LGE): FAS 3
Description: as for outcome 64
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 57
Participants
  Negative | 7
  Positive | 50

66. Secondary Outcome: Number of Participants With Magnetic Resonance Imaging (MRI) Scan Performed Using Late Gadolinium Enhancement (LGE): FAS 3.1
Description: as for outcome 64
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 39
Participants
  Negative | 6
  Positive | 33

67. Secondary Outcome: Number of Participants With Magnetic Resonance Imaging (MRI) Scan Performed Using Late Gadolinium Enhancement (LGE): FAS 3.2
Description: as for outcome 64
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 13
Participants
  Negative | 0
  Positive | 13

68. Secondary Outcome: Number of Participants According to Assessment for Electrocardiogram (ECG) Paced: FAS 2
Description: Participants classified according to assessment for ECG for paced participants as 'Yes' or 'No' were reported in this outcome measure.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 235
Participants
  No | 217
  Yes | 18

69. Secondary Outcome: Number of Participants According to Assessment for Electrocardiogram (ECG) Paced: FAS 3
Description: as for outcome 68
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 200
Participants
  No | 182
  Yes | 18

70. Secondary Outcome: Number of Participants According to Assessment for Electrocardiogram (ECG) Paced: FAS 3.1
Description: as for outcome 68
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 132
Participants
  No | 122
  Yes | 10

71. Secondary Outcome: Number of Participants According to Assessment for Electrocardiogram (ECG) Paced: FAS 3.2
Description: as for outcome 68
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 55
Participants
  No | 49
  Yes | 6

72. Secondary Outcome: Heart Rate Parameter for Participants Without Paced: FAS 2
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | All Participants
Number analyzed (Participants) | 214
Beats per minute | 73.3 (15.1)

73. Secondary Outcome: Heart Rate Parameter for Participants Without Paced: FAS 3
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | All Participants
Number analyzed (Participants) | 179
Beats per minute | 73.2 (14.7)

74. Secondary Outcome: Heart Rate Parameter for Participants Without Paced: FAS 3.1
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | All Participants
Number analyzed (Participants) | 121
Beats per minute | 73.4 (15.9)

75. Secondary Outcome: Heart Rate Parameter for Participants Without Paced: FAS 3.2
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | All Participants
Number analyzed (Participants) | 48
Beats per minute | 72.7 (12.1)

76. Secondary Outcome: Number of Participants Assessed for Sinus Rhythm Parameter for Participants Without Paced: FAS 2
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 227
Participants
  No | 86
  Yes | 135
  Missing | 6

77. Secondary Outcome: Number of Participants Assessed for Sinus Rhythm Parameter for Participants Without Paced: FAS 3
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 190
Participants
  No | 72
  Yes | 114
  Missing | 4

78. Secondary Outcome: Number of Participants Assessed for Sinus Rhythm Parameter for Participants Without Paced: FAS 3.1
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 127
Participants
  No | 51
  Yes | 73
  Missing | 3

79. Secondary Outcome: Number of Participants Assessed for Sinus Rhythm Parameter for Participants Without Paced: FAS 3.2
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 50
Participants
  No | 18
  Yes | 32
  Missing | 0

80. Secondary Outcome: Sokolow Index: FAS 2
Description: Sokolow index is calculated as sum of the amplitude of the S wave in in right precordial lead V1 and the amplitude of the highest R wave in left precordial leads V5 or V6. If the result is greater than 35 mm, it is suggestive of left ventricular hypertrophy.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | All Participants
Number analyzed (Participants) | 180
Millimeter | 19.1 (8.8)

81. Secondary Outcome: Sokolow Index: FAS 3
Description: as for outcome 80
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | All Participants
Number analyzed (Participants) | 148
Millimeter | 18.7 (8.6)

82. Secondary Outcome: Sokolow Index: FAS 3.1
Description: as for outcome 80
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | All Participants
Number analyzed (Participants) | 103
Millimeter | 19.8 (8.7)

83. Secondary Outcome: Sokolow Index: FAS 3.2
Description: as for outcome 80
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | All Participants
Number analyzed (Participants) | 39
Millimeter | 16.5 (8.4)

84. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF): FAS 2
Description: LVEF was defined as the central measure of left ventricular systolic function. LVEF was the fraction of stroke volume (volume ejected in systole) in relation to the volume of the blood in the ventricle at the end of diastole volume (EDV). LVEF was presented in percentage.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percentage of blood volume
Arm/Group | All Participants
Number analyzed (Participants) | 241
Percentage of blood volume | 55.0 (11.4)

85. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF): FAS 3
Description: as for outcome 84
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: Percentage of blood volume
Arm/Group | All Participants
Number analyzed (Participants) | 205
Percentage of blood volume | 55.2 (11.2)

86. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF): FAS 3.1
Description: as for outcome 84
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Percentage of blood volume
Arm/Group | All Participants
Number analyzed (Participants) | 134
Percentage of blood volume | 55.7 (11.2)

87. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF): FAS 3.2
Description: as for outcome 84
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage of blood volume
Arm/Group | All Participants
Number analyzed (Participants) | 56
Percentage of blood volume | 53.9 (11.4)

88. Secondary Outcome: Number of Participants Assessed for Left Ventricular Outflow Tract Obstruction (LVOT): FAS 2
Description: LVOT is defined as limitation of blood flow out of the left ventricle. The level of obstruction can be valvular, sub-valvular, or supravalvular. In this outcome measure participants were categorized as Yes or No on the basis of presence or absence of LVOT.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 241
Participants
  No | 215
  Yes | 26

89. Secondary Outcome: Number of Participants Assessed for Left Ventricular Outflow Tract Obstruction (LVOT): FAS 3
Description: as for outcome 88
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 205
Participants
  No | 183
  Yes | 22

90. Secondary Outcome: Number of Participants Assessed for Left Ventricular Outflow Tract Obstruction (LVOT): FAS 3.1
Description: as for outcome 88
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 136
Participants
  No | 119
  Yes | 17

91. Secondary Outcome: Number of Participants Assessed for Left Ventricular Outflow Tract Obstruction (LVOT): FAS 3.2
Description: as for outcome 88
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 56
Participants
  No | 51
  Yes | 5

92. Secondary Outcome: Number of Participants Categorized According to Perseverance of Strain Apical: FAS 2
Description: Participants were classified according to strain apical preserved as 'No' and 'Yes'.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 90
Participants
  No | 28
  Yes | 62

93. Secondary Outcome: Number of Participants Categorized According to Perseverance of Strain Apical: FAS 3
Description: Participants were classified according to strain apical preserved as 'No' and 'Yes'.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 86
Participants
  No | 26
  Yes | 60

94. Secondary Outcome: Number of Participants Categorized According to Perseverance of Strain Apical: FAS 3.1
Description: Participants were classified according to strain apical preserved as 'No' and 'Yes'.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 62
Participants
  No | 16
  Yes | 46

95. Secondary Outcome: Number of Participants Categorized According to Perseverance of Strain Apical: FAS 3.2
Description: Participants were classified according to strain apical preserved as 'No' and 'Yes'.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 20
Participants
  No | 8
  Yes | 12

96. Secondary Outcome: LV End Diastolic Diameter: FAS 2
Description: Left ventricular end-diastolic diameter (LVEDD) reflects the size of cardiac as well as left ventricular function. It was associated with progressive left ventricular insufficiency.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | All Participants
Number analyzed (Participants) | 218
Millimeter | 43.3 (7.9)

97. Secondary Outcome: LV End Diastolic Diameter: FAS 3
Description: LVEDD reflects the size of cardiac as well as left ventricular function. It was associated with progressive left ventricular insufficiency.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | All Participants
Number analyzed (Participants) | 182
Millimeter | 43.2 (7.9)

98. Secondary Outcome: LV End Diastolic Diameter: FAS 3.1
Description: as for outcome 97
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | All Participants
Number analyzed (Participants) | 120
Millimeter | 43.2 (7.5)

99. Secondary Outcome: LV End Diastolic Diameter: FAS 3.2
Description: as for outcome 97
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | All Participants
Number analyzed (Participants) | 50
Millimeter | 44.4 (6.8)

100. Secondary Outcome: Maximum Wall Thickness: FAS 2
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | All Participants
Number analyzed (Participants) | 240
Millimeter | 17.4 (2.5)

101. Secondary Outcome: Maximum Wall Thickness: FAS 3
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | All Participants
Number analyzed (Participants) | 204
Millimeter | 17.5 (2.4)

102. Secondary Outcome: Maximum Wall Thickness: FAS 3.1
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | All Participants
Number analyzed (Participants) | 136
Millimeter | 17.9 (2.5)

103. Secondary Outcome: Maximum Wall Thickness: FAS 3.2
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | All Participants
Number analyzed (Participants) | 56
Millimeter | 16.9 (2.2)

104. Secondary Outcome: Number of Participants According to Type of Hypertrophic Pattern: FAS 2
Description: Participants were classified according to hypertrophic pattern as apical, concentric, asymmetric and mix.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 240
Participants
  Apical | 6
  Concentric | 179
  Asymmetric | 47
  Mix | 8

105. Secondary Outcome: Number of Participants According to Type of Hypertrophic Pattern: FAS 3
Description: Participants were classified according to hypertrophic pattern as apical, concentric, asymmetric and mix.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 204
Participants
  Apical | 4
  Concentric | 159
  Asymmetric | 37
  Mix | 4

106. Secondary Outcome: Number of Participants According to Type of Hypertrophic Pattern: FAS 3.1
Description: Participants were classified according to hypertrophic pattern as apical, concentric, asymmetric and mix.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 135
Participants
  Apical | 1
  Concentric | 105
  Asymmetric | 27
  Mix | 2

107. Secondary Outcome: Number of Participants According to Type of Hypertrophic Pattern: FAS 3.2
Description: Participants were classified according to hypertrophic pattern as apical, concentric, asymmetric and mix.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 56
Participants
  Apical | 2
  Concentric | 46
  Asymmetric | 7
  Mix | 1

108. Secondary Outcome: LV Mass Index (LVMI): FAS 2
Description: Left ventricular mass (LVM) is the weight of the left ventricle, typically estimated using echocardiography, and is thought to represent the cumulative effect of blood pressure on the heart. Closely related to body size, greater in men than in women, and increases with age. LVMI = LVM (left ventricular mass)/body surface area.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per meter square
Arm/Group | All Participants
Number analyzed (Participants) | 146
Grams per meter square | 172.7 (64.0)

109. Secondary Outcome: LV Mass Index (LVMI): FAS 3
Description: as for outcome 108
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: Grams per meter square
Arm/Group | All Participants
Number analyzed (Participants) | 115
Grams per meter square | 177.0 (53.2)

110. Secondary Outcome: LV Mass Index (LVMI): FAS 3.1
Description: as for outcome 108
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Grams per meter square
Arm/Group | All Participants
Number analyzed (Participants) | 75
Grams per meter square | 177.0 (48.7)

111. Secondary Outcome: LV Mass Index (LVMI): FAS 3.2
Description: as for outcome 108
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Grams per meter square
Arm/Group | All Participants
Number analyzed (Participants) | 31
Grams per meter square | 185.5 (62.0)

112. Secondary Outcome: Aortic Valvular Stenosis - Aortic Valve Area: FAS 2
Description: Aortic valve stenosis is a type of heart valve disease (valvular heart disease). The valve between the lower left heart chamber and the body's main artery (aorta) is narrowed and doesn't open fully. This reduces or blocks blood flow from the heart to the aorta and to the rest of the body. Parameters needed to classify the aortic valve stenosis: peak transvalvular velocity, mean pressure gradient and aortic valve area. Here, aortic valve area is reported in this outcome measure.
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Centimeter square
Arm/Group | All Participants
Number analyzed (Participants) | 146
Centimeter square | 2.3 (0.8)

113. Secondary Outcome: Aortic Valvular Stenosis - Aortic Valve Area: FAS 3
Description: as for outcome 112
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: Centimeter square
Arm/Group | All Participants
Number analyzed (Participants) | 123
Centimeter square | 2.2 (0.7)

114. Secondary Outcome: Aortic Valvular Stenosis - Aortic Valve Area: FAS 3.1
Description: as for outcome 112
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Centimeter square
Arm/Group | All Participants
Number analyzed (Participants) | 83
Centimeter square | 2.3 (0.7)

115. Secondary Outcome: Aortic Valvular Stenosis - Aortic Valve Area: FAS 3.2
Description: as for outcome 112
Time Frame: During collection and observation duration from 09-Jul-2018 to 08-Jun-2022 (approximately 3.11 years)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Centimeter square
Arm/Group | All Participants
Number analyzed (Participants) | 34
Centimeter square | 2.0 (0.7)

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not planned to be collected during the study
Description: Minimum criteria for reporting an adverse event (i.e. identifiable participant, identifiable reporter, a suspect product, and event) could not be met. Hence, adverse events were not collected and reported.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT03842163/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT03842163/SAP_001.pdf